CLINICAL TRIAL: NCT02347787
Title: A Multi-center Trial of Clinician Versus Community Health Worker Support to Help Low Socioeconomic, Chronically-ill Patients Achieve Health Goals
Brief Title: A Multi-center Trial of IMPaCT CHW Support for Chronically-ill Patients
Acronym: IMPaCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 821368
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Diabetes; Obesity; Tobacco Dependence
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Obesity; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual clinician support (Placebo Comparator): Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the usual clinician support arm will receive usual care in accordance with guidelines at each site.
  Interventions: Other: Usual care
- CHW support (Experimental): Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the CHW arm will receive the IMPaCT intervention.
  Interventions: Behavioral: IMPaCT

INTERVENTIONS:
Behavioral: IMPaCT — The IMPaCT intervention has three stages:
  1. Goal-setting: CHWs will help patients to deconstruct the chronic disease management goal they set with their PCP into patient-driven short-term goals and action plans.
  2. Tailored Support: CHWs will conduct weekly follow-up for 6 months through either telephone or home visit in order to support the achievement of patients' short-term goals.
  3. Connection with longitudinal support: IMPaCT CHWs will also facilitate a weekly patient support group.
  Arms: CHW support
Other: Usual care
  Arms: Usual clinician support

SUMMARY:
This is a multi-center randomized controlled trial comparing the effectiveness of community health worker (CHW) vs. usual clinician support in helping chronically-ill patients with low socioeconomic status to improve their health outcomes.

DETAILED DESCRIPTION:
Community Health Workers (CHWs) have the potential to improve chronic disease outcomes among patients with low socioeconomic status (SES). Yet, widespread use of CHWs has been hampered by lack of standardized, scalable and evidence-based models. Our community-academic-health system team used participatory action research with low-SES patients to design IMPaCT (Individualized Management for Patient-Centered Targets). A randomized controlled trial (RCT) of 446 hospitalized patients with varied diseases demonstrated that a 2-week dose of IMPaCT improved access to care, mental health, activation, and quality of communication, while reducing recurrent hospital readmissions. We have adapted IMPaCT for use among low-SES primary care patients with multiple chronic conditions.

This RCT is designed to evaluate the newly adapted IMPaCT model in 3 primary care settings - academic, federally qualified health center, and VA. Upon enrollment in the trial, patients will collaboratively set a chronic disease management goal with their primary care provider. Patients will then be randomized to collaborative goal-setting versus goal-setting augmented by 6 months of support from an IMPaCT CHW. Follow-up will be conducted at 6- and 9- months post-enrollment.

The study design is a single-blinded, 2- armed, multi-site randomized controlled trial involving three clinic sites and 444 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient of specific practice (Mutch/St.Leonards Court, Spectrum, PVAMC) for at least 1 yr defined as having one office visit within preceding 12 months
* Resident of home ZIP code including ANY of the following 19104, 19131, 19139, 19142, 19143, 19145, 19146, & 19151
* Has 2 or more of the following conditions: 1. Obesity: BMI30 2. HTN: ICD9 relating to HTN from EMR problem list or EMR ICD9 encounter diagnosis x2) 3.DM: ICD9 relating to DM from EMR problem list or EMR ICD9 encounter diagnosis x2) 4. tobacco (from EPIC Social History/Vital Signs)
* Has at least one poorly controlled condition based on the most recent value prior to enrollment: Obesity (BMI>=35); HTN (SBP >= 160); DM (HgBA1c >=9); Tobacco Use (>0 cigarettes)"
* Is uninsured, insured by Medicaid, or dually eligible for Medicare and Medicaid or VA Insurance
* Has a scheduled appointment at a study clinic in the future.
* Community Health Workers/CHWs/IMPaCT Partners involved in the care of patients of the three practices will be included in the qualitative portion of this study.

Exclusion Criteria:

* Will not provide informed consent for this study.
* Does not have the capacity to provide informed consent for this study.
* Previously enrolled in this study.
* Currently enrolled in another study focusing on chronic disease management.
* Currently has a CHW
* No one will be excluded on the basis of sex or race.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Long, MD, Principal Investigator — University of Pennsylvania/Philadelphia Veterans Affairs Medical Center

REFERENCES:
- [Derived] Kangovi S, Mitra N, Norton L, Harte R, Zhao X, Carter T, Grande D, Long JA. Effect of Community Health Worker Support on Clinical Outcomes of Low-Income Patients Across Primary Care Facilities: A Randomized Clinical Trial. JAMA Intern Med. 2018 Dec 1;178(12):1635-1643. doi: 10.1001/jamainternmed.2018.4630. PMID 30422224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment took place at: a Veterans Affairs medical center primary care practice, a federally qualified health center and an academic family medicine clinic. Patients were recruited between January 28th, 2015 and March 28, 2016 at which time the trial was stopped because we had reached our pre-specified sample size target.
Groups:
- Usual Clinician Support: Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the usual clinician support arm will receive usual care in accordance with guidelines at each site.
  Usual care
- CHW Support: Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the CHW arm will receive the IMPaCT intervention.
  IMPaCT: The IMPaCT intervention has three stages:
  1. Goal-setting: CHWs will help patients to deconstruct the chronic disease management goal they set with their PCP into patient-driven short-term goals and action plans.
  2. Tailored Support: CHWs will conduct weekly follow-up for 6 months through either telephone or home visit in order to support the achievement of patients' short-term goals.
  3. Connection with longitudinal support: IMPaCT CHWs will also facilitate a weekly patient support group.
Period: 6 Month Follow-Up
Arm/Group | Usual Clinician Support | CHW Support
Started | 288 | 304
Completed | 222 | 248
Not Completed | 66 | 56
Not completed — Lost to Follow-up | 63 | 47
Not completed — Withdrawal by Subject | 3 | 9
Period: 9 Month Follow-Up
Arm/Group | Usual Clinician Support | CHW Support
Started | 288 | 304
Completed | 227 | 233
Not Completed | 61 | 71
Not completed — Lost to Follow-up | 52 | 59
Not completed — Withdrawal by Subject | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Clinician Support | CHW Support | Total
Number analyzed (Participants) | 288 | 304 | 592
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.5) | 53.1 (10.7) | 52.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 194 | 370
  Male | 112 | 110 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 11 | 11
  Not Hispanic or Latino | 285 | 285 | 570
  Unknown or Not Reported | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 274 | 284 | 558
Employed [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 286 | 303 | 589
    (all) | 48 | 47 | 95
Household Income [Count of Participants; unit: Participants]
  < 15K | 186 | 197 | 383
  > 15K | 69 | 69 | 138
  Unknown | 33 | 38 | 71
Trauma History [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 286 | 304 | 590
    (all) | 280 | 297 | 577
Low Social Support [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 286 | 304 | 590
    (all) | 57 | 76 | 133
Short Grit Scale (Grit-S) [Mean (Standard Deviation); unit: units on a scale] — This scale asks 8 questions relating to a person's passion and perseverance. Each question is graded on a five point likert scale where respondents rate statements as being somewhere from 'Not like me at all' to 'Very much like me'. Scores from each of the 8 questions are averaged for a total grit score with 5 being high grit (high passion/perseverance) and 1 being low grit. Population: Not all participants answered this question.
  units on a scale
    number analyzed (Participants) | 285 | 304 | 589
    (all) | 2.7 (0.5) | 2.7 (0.6) | 2.7 (0.5)
Adult Attachment Questionnaire (AAQ) [Mean (Standard Deviation); unit: units on a scale] — The Adult Attachment Questionnaire (AAQ) is an 11-item scale that measures secure, avoidant, and anxious attachment styles. For each question, the participant is asked to rate a statement on a scale of 1-6 (Strongly agree, agree, slightly agree, slightly disagree, disagree, strongly disagree). Scores are then averaged to get a final score between 1 and 6.
  Some of the questions can be combined to create subscores for avoidance and anxiety. Higher scores on these dimensions reflect greater avoidance or anxiety. Greater attachment security is defined by lower scores on both scales.
  units on a scale
    Secure | 3.4 (0.9) | 3.4 (0.9) | 3.4 (0.9)
    Avoidant | 3.6 (1.3) | 3.7 (1.3) | 3.6 (1.3)
    Anxious | 2.9 (1.8) | 2.8 (1.8) | 2.9 (1.8)
Delayed Health Need [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 283 | 302 | 585
    (all) | 129 | 143 | 272
Unmet health Need [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 283 | 303 | 586
    (all) | 81 | 76 | 157
Lack of Basic needs [Count of Participants; unit: Participants] | 118 | 120 | 238
Alcohol Overuse [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 259 | 272 | 531
    (all) | 73 | 81 | 154
Drug Use [Count of Participants; unit: Participants] — Population: Not all participants answered this question.
  Participants
    number analyzed (Participants) | 283 | 303 | 586
    (all) | 69 | 63 | 132
Short Form Health Survey (SF-12) [Mean (Standard Deviation); unit: score on a scale] — The SF-12 is a survey designed for use with patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5 point likert scale and 2 are answered on a 3 point likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health. A 3 point change in SF-12 score reflects a meaningful difference. Population: Not all participants answered these questions.
  score on a scale
    Mental Health Component: number analyzed (Participants) | 286 | 304 | 590
    Mental Health Component | 43.1 (12.9) | 42.2 (14.1) | 42.7 (13.5)
    Physical Health Component: number analyzed (Participants) | 286 | 304 | 590
    Physical Health Component | 33.6 (9.9) | 34.0 (10.7) | 33.8 (10.3)
Patient Activation Measure (PAM) [Mean (Standard Deviation); unit: units on a scale] — The PAM is a 13-item survey that assesses a person's underlying knowledge, skills, and confidence integral to managing his or her own health and healthcare. Respondents are asked to strongly agree, agree, disagree, or strongly disagree with each statement. Responses are then scored into a 100 point scale where higher scores indicate increased patient activation (higher knowledge, skills, and confidence for managing their own health/healthcare). Population: Not all participants answered these questions.
  units on a scale
    number analyzed (Participants) | 286 | 304 | 590
    (all) | 60.8 (14.3) | 59.4 (14.2) | 60.1 (14.3)
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — The PSS measures how much stress a person attributes to various situations in their life. While the PSS is a 10 point scale, a short form of 4 questions was used for this study. Each question on the scale is rated from Never (0) to Very Often (4). Scores are then summed. For the 4 question short form there is a range of scores between 0 and 16 with 16 being the highest level of stress and 0 being no stress. Population: Not all participants answered these questions.
  units on a scale
    number analyzed (Participants) | 286 | 304 | 590
    (all) | 6.7 (3.3) | 6.7 (3.5) | 6.7 (3.4)
Single Item Literacy Screener (SILS) [Mean (Standard Deviation); unit: units on a scale] — This single item screener assesses how much assistance respondents need in reading health-related materials. This is scored as a 5 point likert scale with a range of 1 - 5. A lower score on this scale indicates high health literacy (never or rarely needing assistance reading health-related materials). A higher score indicates low health literacy (often or always needing assistance reading health-related materials). Population: Not all participants answered this question.
  units on a scale
    number analyzed (Participants) | 286 | 304 | 590
    (all) | 1.9 (1.1) | 2.1 (1.3) | 2.0 (1.2)
ER visits in prior 12 months [Mean (Standard Deviation); unit: Avg # of visits] | 2.2 (3.5) | 1.8 (2.1) | 2.0 (2.9)
Admissions in prior 12 months [Mean (Standard Deviation); unit: Avg # of admissions] | 1.0 (2.5) | 0.7 (1.1) | 0.9 (1.9)
Chronic Disease Prevalence - Hypertension [Count of Participants; unit: Participants] | 257 | 263 | 520
Chronic Disease Prevalence - Obesity [Count of Participants; unit: Participants] | 228 | 240 | 468
Chronic Disease Prevalence - Diabetes [Count of Participants; unit: Participants] | 134 | 139 | 273
Chronic Disease Prevalence - Tobacco Dependence [Count of Participants; unit: Participants] | 104 | 124 | 228
Selected Condition [Count of Participants; unit: Participants]
  Hypertension | 33 | 30 | 63
  Obesity | 149 | 157 | 306
  Diabetes | 35 | 34 | 69
  Tobacco Dependence | 71 | 83 | 154
Hypertension [Mean (Standard Deviation); unit: mmHg] — Baseline clinical parameters and health goal among those participants who focused on a hypertension reduction goal. To measure this outcome, we are assessing systolic blood pressure values in mmHg Population: Each participant was asked to focus on one chronic condition to set a health goal for the study. Because of this, the number of participants analyzed for this outcome is less than the overall number of participants in the study.
  mmHg
    Baseline Control: number analyzed (Participants) | 33 | 30 | 63
    Baseline Control | 159.8 (26.5) | 163.4 (19.3) | 161.6 (23.3)
    Hypertension Goal: number analyzed (Participants) | 33 | 30 | 63
    Hypertension Goal | -26.4 (34.6) | -24.1 (17.9) | -25.3 (27.7)
Diabetes [Mean (Standard Deviation); unit: HbA1c%] — Baseline clinical parameters and collaboratively set health goal among those participants who focused on a diabetes goal. Patients were asked to set a goal with their health care provider to lower their Hemoglobin A1c. Population: Each participant was asked to focus on one chronic condition to set a health goal for the study. Because of this, the number of participants analyzed for this outcome is less than the overall number of participants in the study.
  HbA1c%
    Baseline Control: number analyzed (Participants) | 35 | 34 | 69
    Baseline Control | 10.5 (2.0) | 10.5 (2.0) | 10.5 (2.0)
    Diabetes Goal: number analyzed (Participants) | 35 | 34 | 69
    Diabetes Goal | -2.3 (1.8) | -2.3 (2.2) | -2.3 (2.0)
Obesity - Baseline Clinical Parameters [Mean (Standard Deviation); unit: kg/m^2 (BMI)] — Baseline clinical parameters among those participants who focused on an obesity reduction goal. Population: Each participant was asked to focus on one chronic condition to set a health goal for the study. Because of this, the number of participants analyzed for this outcome is less than the overall number of participants in the study.
  kg/m^2 (BMI)
    number analyzed (Participants) | 149 | 157 | 306
    (all) | 42.2 (6.9) | 42.8 (8.1) | 42.5 (7.5)
Obesity - Health Goal [Mean (Standard Deviation); unit: pounds] — Collaboratively set health goal among those participants who focused on an obesity reduction goal. Patients were asked to set a goal with their health care provider to lower their BMI. The goal was set in pounds. Population: Each participant was asked to focus on one chronic condition to set a health goal for the study. Because of this, the number of participants analyzed for this outcome is less than the overall number of participants in the study.
  pounds
    number analyzed (Participants) | 149 | 157 | 306
    (all) | -15.1 (5.6) | -14.7 (6.3) | -14.9 (6.0)
Tobacco Use [Mean (Standard Deviation); unit: number of cigarettes] — Baseline number of cigarettes smoked per day among those participants who focused on a tobacco cessation goal. This was measured by self-reported daily tobacco use ("How many cigarettes do you smoke a day?"). All participants who focused on tobacco use were asked to set a quit smoking goal so there is no collaboratively set goal indicator for this chronic disease outcome. Population: Each participant was asked to focus on one chronic condition to set a health goal for the study. Because of this, the number of participants analyzed for this outcome is less than the overall number of participants in the study.
  number of cigarettes
    number analyzed (Participants) | 71 | 83 | 154
    (all) | 9.7 (7.2) | 8.9 (6.4) | 9.3 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Short Form Health Survey (SF-12) Physical Component Score (PCS)
Description: The main dependent variable is mean change in standardized score for SF-12 PCS. The SF-12 is a survey designed for use with patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5 point likert scale and 2 are answered on a 3 point likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health. A 3 point change in SF-12 score reflects a meaningful difference. We measure the between-arm difference in mean change in SF-12 PCS between baseline and 6-month follow-up assessment.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinician Support | CHW Support
Number analyzed (Participants) | 222 | 248
score on a scale | 2.3 (11.3) | 0.6 (12.7)
Statistical Analysis 1: Comparison: Usual Clinician Support vs CHW Support; Determination of targeted sample size was based on detecting a between-arm difference in mean change in SF-12 Physical Component Summary of 3 points, which is the minimal clinically significant difference for this instrument. To achieve at least 80% power with a type I error rate of 5%, we required 444 total participants. To account for 25% attrition, we aimed to accrue 592 participants; Test type: Superiority; p = 0.30, Regression, Linear

2. Secondary Outcome: Change in Chronic Disease Control - Diabetes
Description: We will asses change in chronic disease control using biometric testing (HgA1c). At six months after enrollment, all patients underwent a clinic visit and the appropriate laboratory testing: HgbA1c. Patients' measurements on this parameter will be used to determine their change in standardized score for their outcome of interest.
Time Frame: Baseline, 6 months, 9 months
Population: Each participant was only analyzed for their chosen chronic condition.
Measure: Mean (Standard Deviation); unit: HbA1c%
Groups:
- Usual Clinician Support - 6 Months; Usual Clinician Support - 9 Months: Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the usual clinician support arm will receive usual care in accordance with guidelines at each site.
  Usual care
- CHW Support - 6 Months; CHW Support - 9 Months: Prior to randomization, patients in this arm will already have set a chronic disease management goal with their primary care provider (who will have received training in collaborative goal-setting). After randomization, patients in the CHW arm will receive the IMPaCT intervention.
  IMPaCT: The IMPaCT intervention has three stages:
  1. Goal-setting: CHWs will help patients to deconstruct the chronic disease management goal they set with their PCP into patient-driven short-term goals and action plans.
  2. Tailored Support: CHWs will conduct weekly follow-up for 6 months through either telephone or home visit in order to support the achievement of patients' short-term goals.
  3. Connection with longitudinal support: IMPaCT CHWs will also facilitate a weekly patient support group.
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 29 | 27 | 29 | 23
HbA1c% | -6.5 (26.0) | -10.9 (16.3) | -10.4 (22.5) | -17.9 (19.5)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.21, Regression, Linear; Risk Difference (RD) = -0.2, 95% CI 2-sided [-1.3 to 0.9]

3. Secondary Outcome: Change in Chronic Disease Control - Obesity
Description: We will asses change in chronic disease control using biometric testing (kg/m^2). At six and nine months after enrollment, all patients underwent a clinic visit and the appropriate laboratory testing: height and weight. Patients' measurements on this parameter will be used to determine their change in standardized score for their outcome of interest.
Time Frame: Baseline, 6 months, 9 months
Population: Each participant was only analyzed for their chosen chronic condition.
Measure: Mean (Standard Deviation); unit: kg/m^2 (BMI)
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 118 | 135 | 120 | 120
kg/m^2 (BMI) | -0.3 (2.5) | -0.5 (2.3) | -0.4 (2.7) | -0.5 (3.0)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.21, Regression, Linear; Risk Difference (RD) = -0.2, 95% CI 2-sided [-0.7 to 0.4]

4. Secondary Outcome: Change in Chronic Disease Control - Tobacco Use
Description: We will asses change in chronic disease control using patient self-report (cigarettes per day). At six and nine months after enrollment, all patients underwent a clinic visit and the appropriate laboratory testing. Patients' measurements on this parameter will be used to determine their change in standardized score for their outcome of interest.
Time Frame: Baseline, 6 months, 9 months
Population: Each participant was only analyzed for their chosen chronic condition.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 52 | 68 | 48 | 67
cigarettes per day | -3.1 (7.1) | -3.5 (6.4) | -3.5 (6.5) | -4.1 (5.4)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.21, Regression, Linear; Risk Difference (RD) = -0.5, 95% CI 2-sided [-2.2 to 1.2]

5. Secondary Outcome: Change in Chronic Disease Control - Hypertension
Description: We will asses change in chronic disease control using biometric testing (systolic blood pressure in mm Hg). At six and nine months after enrollment, all patients underwent a clinic visit and the appropriate laboratory testing. Patients' measurements on this parameter will be used to determine their change in standardized score for their outcome of interest.
Time Frame: Baseline, 6 months, 9 months
Population: Each participant was only analyzed for their chosen chronic condition.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 29 | 27 | 29 | 23
mm Hg | -6.2 (26.0) | -10.9 (16.3) | -10.4 (22.5) | -17.9 (19.5)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.21, Regression, Linear; Risk Difference (RD) = -6.3, 95% CI 2-sided [-14.3 to 1.8]

6. Secondary Outcome: Short Form Health Survey (SF-12) - Mental Component Summary (MCS)
Description: The SF-12 is a survey designed for use with patients with multiple chronic conditions. This 12-item scale can be used to assess the physical and mental health of respondents. 10 of the 12 questions are answered on a 5 point likert scale and 2 are answered on a 3 point likert scale. The questions are then scored and weighted into 2 subscales, physical health and mental health. Respondents can have a score that ranges from 0-100 with 100 being the best score and indicating high physical or mental health. A 3 point change in SF-12 score reflects a meaningful difference. We will assess this outcome using the SF-12 Mental Component Summary (MCS) score. The MCS reliably detects differences in mental health over time. We will measure the between-arm difference in mean change in SF-12 MCS score between baseline, 6- and 9- month follow-up.
Time Frame: Baseline, 6 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 222 | 248 | 227 | 233
score on a scale | 1.7 (14.1) | 2.2 (13.3) | 1.2 (13.7) | 2.2 (14.1)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.41, Regression, Linear

7. Secondary Outcome: Number of Participants Reporting Highest Rating for Quality of Patient-centered Care - Comprehensiveness
Description: We will assess this outcome using the Consumer Assessment of Healthcare Providers and Systems Patient-Centered Medical Home (CAHPS PCMH) survey. This survey assesses the quality of patient-centered primary care and can be used by any practice (not just PCMH practices). We will measure the CAHPS PCMH domains pertaining to Self-Management Support and Comprehensiveness of Care. We will measure the number of patients who gave the highest rating of care for the comprehensiveness question at 6 and 9 months post-enrollment.
Time Frame: 6 months, 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 222 | 248 | 227 | 233
Participants | 83 | 137 | 97 | 139
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p < 0.001, Regression, Logistic

8. Secondary Outcome: Number of Participants With Any Hospital Admission
Description: We will measure admission to hospital at 6- and 9 months after enrollment. This data will be obtained through 1) self-report, 2) the Pennsylvania Cost Containment Council (PHC4), a state-based initiative that tracks utilization data across the state of Pennsylvania, 3) the Veterans Affairs electronic medical record, 4) the Penn electronic medical record
Time Frame: 6 months and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 222 | 248 | 227 | 233
Participants | 35 | 38 | 51 | 52
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.98, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.5]

9. Secondary Outcome: Qualitative Assessment of Intervention and Mechanisms Affecting Achievement of Primary Outcome
Description: At 6-months post-enrollment, a trained qualitative interviewer on our study team will conduct an in-depth qualitative semi-structured interview with 40 intervention arm patients and their CHWs. Qualitative interviews will be audio-taped and transcribed. Patients will be purposively sampled across each study site in order to be able to make comparisons between those who achieved a minimally important improvement in the primary outcome and those who did not. These interviews will be guided by the Integrative Behavior Model (IBM). UPDATE: After beginning interviews, our team decided that 26 interviews was sufficient to reach thematic saturation.
Time Frame: 6 months
Population: This data point contains qualitative, not quantitative data. The study team is still analyzing this data set and has not yet completed analysis for this outcome. Below, we report the number of interviews completed for each clinical site (VA, Federally Qualified Health Center, Academic Site). We will not complete any more interviews.
Measure: Count of Participants; unit: Participants
Arm/Group | CHW Support
Number analyzed (Participants) | 26
Participants
  VA | 10
  FQHC | 10
  Academic Site | 6

10. Secondary Outcome: Number of Participants Reporting the Highest Rating for Quality of Patient-centered Care - Supportiveness of Self-management
Description: We will assess this outcome using the Consumer Assessment of Healthcare Providers and Systems Patient-Centered Medical Home (CAHPS PCMH) survey. This survey assesses the quality of patient-centered primary care and can be used by any practice (not just PCMH practices). We will measure the CAHPS PCMH domains pertaining to Self-Management Support and Comprehensiveness of Care. We will measure the number of patients who gave the highest rating of care for the supportiveness of disease self-management question at 6 and 9 months post-enrollment.
Time Frame: 6 months, 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 222 | 248 | 227 | 233
Participants | 95 | 157 | 112 | 145
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p < 0.001, Regression, Logistic

11. Secondary Outcome: Number of Participants With Multiple Hospital Admissions
Description: as for outcome 8
Time Frame: 6 months and 9 months
Population: This outcome was only assessed for participants who had hospital admission. Therefore the number of participants analyzed is smaller than that for the overall study.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 35 | 38 | 51 | 52
Participants | 14 | 4 | 21 | 15
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.02, Regression, Logistic

12. Secondary Outcome: Number of Participants With 30 Day Hospital Readmissions
Description: We will measure admission to hospital at 30 days after enrollment. This data will be obtained through 1) self-report, 2) the Pennsylvania Cost Containment Council (PHC4), a state-based initiative that tracks utilization data across the state of Pennsylvania, 3) the Veterans Affairs electronic medical record, 4) the Penn electronic medical record
Time Frame: 30 days
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 35 | 38 | 51 | 52
Participants | 9 | 3 | 14 | 6
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.04, Regression, Logistic

13. Secondary Outcome: Hospital Admission - Total Hospital Days
Description: as for outcome 8
Time Frame: 6 months and 9 months
Measure: Number; unit: Days
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 288 | 304 | 288 | 304
Days | 345 | 155 | 471 | 300

14. Secondary Outcome: Hospital Admission - Mean Number of Hospitalizations
Description: as for outcome 8
Time Frame: 6 months and 9 months
Population: This outcome was only assessed for participants who had a hospital admission. Therefore the number of participants analyzed is smaller than that for the overall study.
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 35 | 38 | 51 | 52
Hospitalizations | 1.5 (0.7) | 1.1 (0.4) | 1.6 (1.0) | 1.4 (0.8)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.09, Regression, Linear

15. Secondary Outcome: Hospital Admission - Mean Length of Stay (Among Participants With Hospitalization)
Description: as for outcome 8
Time Frame: 6 months and 9 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Clinician Support - 6 Months | CHW Support - 6 Months | Usual Clinician Support - 9 Months | CHW Support - 9 Months
Number analyzed (Participants) | 35 | 38 | 51 | 52
days | 9.9 (17.5) | 4.1 (3.1) | 9.2 (15.3) | 5.8 (6.5)
Statistical Analysis 1: Comparison: Usual Clinician Support - 6 Months vs CHW Support - 6 Months vs Usual Clinician Support - 9 Months vs CHW Support - 9 Months; Test type: Superiority; p = 0.06, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months when participants were actively working on their chronic disease management goals. We did not collect or monitor any adverse event data after 6 months as participants were no longer engaged with a CHW/working on their health goals at that time.
Arm/Group | Usual Clinician Support | CHW Support
All-Cause Mortality (participants affected / at risk) | 3/288 | 1/304
Serious Adverse Events (participants affected / at risk) | 32/288 | 35/304
Other Adverse Events (participants affected / at risk) | 0/288 | 0/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Clinician Support (N=288) | CHW Support (N=304)
Blood infection (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Allergic reaction to meds (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Angioplasty (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (6)
Bowel Issues (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bacterial Infection (Infections and infestations) | 1 (1) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Injuries due to fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gynecological Issues (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Diabetes Complications (Endocrine disorders) | 1 (1) | 3 (3)
Blood Pressure Issues (Blood and lymphatic system disorders) | 1 (2) | 4 (4)
Kidney Issues (Renal and urinary disorders) | 2 (2) | 1 (1)
Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Swelling and pain in lower extremities (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Death - Cause Unknown (General disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pregnancy Complications (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 1 (1)
Stroke (Vascular disorders) | 5 (5) | 1 (1)
Ulcers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dog Bite (Social circumstances) | 0 (0) | 1 (1)
Skin wound (General disorders) | 0 (0) | 1 (1)
Gallstones (Renal and urinary disorders) | 0 (0) | 1 (1)
Heart Attack (Vascular disorders) | 0 (0) | 1 (1)
Hernia Repair (General disorders) | 0 (0) | 2 (2)
Hit by a car (Social circumstances) | 0 (0) | 1 (1)
Inpatient Psych Evaluation (Social circumstances) | 0 (0) | 1 (1)
(General disorders) | 0 (0) | 1 (1)
Respiratory Issues (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dehydration (Social circumstances) | 0 (0) | 1 (1)
Blood Transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No